CLINICAL TRIAL: NCT04038736
Title: Evaluation of Check-Cap C-Scan System in Providing Structural Information and Detection of Polypoid Lesions in Subjects at Average or High Risk for CRC
Brief Title: Evaluation C-Scan System in Providing Structural Information and Polypoid Lesions in the Colon of Healthy Subjects
Acronym: CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CL-SY-01-0098
Record Dates: First submitted 2019-06-27; First posted 2019-07-31 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Risk for Colorectal Cancer

STUDY DESIGN:
Intervention Model Description: Evaluation of the performance of the C-Scan System in providing structural information on colonic polypoid lesions and masses in average risk vs. high risk subjects.
Who Masked: Outcomes Assessor
Masking Description: 3 independent reviewers, licensed physicians, trained with reviewing and analyzing C-Scan System scans, will evaluate all study subjects original scans for potential findings, including type, location and size. All reviewers will be blinded to the subject groups (symptoms, classification etc.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects at averge risk for CRC (Experimental): All subjects are healthy who didn't have any known polyps in past colonoscopy and who arw candidates for CRC screening
  Interventions: Device: C-Scan System
- Healthy subjects at high risk for CRC (Experimental): Subjects who had polyps in former colonoscopy, subjects who have family history of CRC or subjects who have positive stool blood test.
  Interventions: Device: C-Scan System

INTERVENTIONS:
Device: C-Scan System — During C-Scan procedure the subject swallows the C-Scan cap. The capsule travels painlessly through the gastrointestinal tract, seeking polyps, the precursors of colorectal cancer. It is essential to increase the stool's contrast by ingesting radio-opaque material. During the passage of the capsule in the gastrointestinal tract, it transmits information to a recorder attached to the back. In order to collect data about the instantaneous localization of the capsule traveling in the colon additional sensors are embedded in the recorder on the back side. After the capsule is expelled, the data from the recorder is downloaded to an acquisition workstation. Later, the data is transferred to a processing workstation where dedicated software visualizes and analyses the data.
  Other Names: C-Scan Cap, C-Scan Track

SUMMARY:
Up to 300 subjects will participate in this study. Subjects to be enrolled in this study are typically healthy and at average or high risk for CRC.

Each subject will undergo study assessments including a pre-screening telephone call, Procedure Visit, follow up post-ingestion via telephone calls.

On the day of the procedure, before administering the C-Scan. Once informed consent is obtained, a thorough evaluation of subject's eligibility will be performed based on inclusion / exclusion criteria. Medical history and concomitant medications information will be collected for all subjects. Also prior surgeries or endoscopic examinations showing pathology and current or previous GI problems or symptoms will be evaluated.

Some subjects will be asked to participate in additional ingestions (up to three, one at a time, at least one week intermission between the ingestions), to compare the performance of the system in different configuration on the same subject.

Each subject's participation in the study will take up to 3 weeks (per one ingestion).

Some subjects will be asked to participate in addition ingestions (up to three, one at a time, at least one week intermission between the ingestions), to compare the performance of the system in different configuration on the same subject.

Overall study duration will be one year.

DETAILED DESCRIPTION:
Study Population:

A total of 300 healthy subjects, Male or female, at average or high risk for CRC will be enrolled for the study.

Visit 1: C-Scan Procedure Visit This visit is performed in order to ensure that the subject continues to meet all inclusion and has no exclusion criteria, and has had adequate time to review the consent form and to ask questions. Once it has been determined that the subject meets all inclusion and has no exclusion criteria, and the subject chooses to participate in the study, the consent form will be signed and dated by all appropriate parties prior to execution of study-specific assessments. Signing the informed consent form signifies enrollment in the clinical study.

Capsule ingestion will take place at this visit. Additionally, the subject will receive detailed training session and instructions including explanation from the site study team about the device, its usage and the required documentation described below. Following subject training, the Capsule will be ingested ('C-Scan Initiation Procedure') at this visit, as described below.

C-Scan Initiation Procedure:

Subject will be connected to the C-Scan Track and system will be activated. The subject will be asked to ingest the C-Scan Capsule, in the presence of a physician with some water and water-soluble iodinated oral contrast medium indicated for radiographic examination of segments of the gastrointestinal tract and non-soluble fiber supplements.

Post ingestion, the subject will be discharged home with a Subject Instructions Packet which will include instructions on following routine daily regime (i.e., ingestion of contrast media 3 x 15ml per day and non-soluble fiber supplements X3 per day until capsule excretion) and record in a personal formatted diary the timing of specific activities such as bowel movements, daily activities and discomfort assessment via a validated scale. Also included will be Subject Satisfaction surveys that the subject should complete at the end of the procedure and return to the site upon completion.

Capsule Progress Days:

During the days in which the capsule is progressing within the subject, the subject is required to ingest contrast media (GE Omnipaque 350, FDA approved under NDA 018956) as well as non-soluble fiber supplements. The subject will be required to ingest daily dose (3 X 15 ml) of contrast media, to be consumed three times per day as well a non-soluble fiber 3x/day with normal diet.

Subjects will be required to undergo FIT procedure along with the C-Scan System procedure, per package insert instructions The subject will be provided with Laxadin (5 mg tablets) to be ingested according to the doctor recommendation, on an as needed basis. In routine procedures, subjects might be instructed to take 2 X 5 mg tablets 48-72 hours after ingestions (unless the capsule was already excreted).

Some subjects will be asked by the PI to come to the site for an abdominal X-Ray (fluoroscopy) while the capsule is still in the colon.

All subjects will be required to keep a log ('Subject's Diary') during procedure documenting general activities, contrast media intake, fibers intake, and food consumption, bowel movement, and system visual/auditory indicators.

Phone Call Follow-Up During-C-Scan Procedure :

After Capsule ingestion, the subject will be contacted by phone at least twice daily by the study team until the capsule has been excreted. The subject will be asked to provide feedback about the use of the device, excretion of the capsule, his/her general feeling or any inconvenience and will be reminded to complete the daily diary and discomfort assessment. The conversation with the subjects and their responses are tabulated and recorded in the study file.

C-Scan Procedure End:

Capsule procedure is completed upon capsule excretion or system auditory indication of 'End of Procedure'. Subjects will be asked to call the study team upon capsule excretion.

The subjects will be provided with a dedicated capsule collection kit, to assist the subjects in collecting the capsule. Subjects will be instructed to retrieve the capsule upon excretion. Return packaging and instructions will be provided. The subject will return with the Kit the diary, the questionnaire and all unused materials.

Follow-Up Phone Call Post-C-Scan Procedure End:

Follow up window is 1-3 days post-capsule excretion. Subject will be telephoned by study site to assess for any undesired events.

In case of doubt regarding capsule excretion, and per physician discretion, subjects may be referred to abdominal X-Ray to confirm capsule excretion.

Colonoscopy examination (optional)

ELIGIBILITY:
Inclusion Criteria:

* Male or female at the age of 40-80 years old
* Subjects who are ready to undergo the monitoring routine
* Subject provided signed informed consent

Exclusion Criteria:

* Subjects with advanced cancer or other life threatening diseases or conditions
* Subjects with known history of dysphagia or other swallowing disorders
* Subjecta with known history of GI disease or symptoms, such as: Crohn's disease, Colitis, IBD, Meckel's Diverticulum, Bowen Hernia, Mega Colon, fistulas or other strictures (doctors' discretion).
* Subject with known motility disorder or Chronic Constipation (less than 3 bowel movements/week)
* Subject with known delayed gastric emptying
* Subjects with prior history of abdominal surgery that might cause bowel strictures leading to capsule retention, as determined by physician discretion
* Subject with any condition believed to have an increased risk for capsule retention such as intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or NSAID enteropathy, as determined by physician discretion
* Subject with a cardiac pacemaker or other implanted electro medical device
* Subjects with known sensitivity to iodine, or with kidney failure
* Subjects with low BMI (BMI<20) or Obese (BMI≥ 38)
* Subjects with belly / girth circumference > 125 cm
* Subject with any known condition which precludes compliance with study and/or device instructions
* Subject with known condition of drug abuse and/or alcoholism
* Women who are either pregnant or nursing at the time of screening (to be verified by test in case of woman of child-bearing potential that do not practice medically acceptable methods of contraception)
* Concurrent participation in another clinical trial using any investigational drug or device

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2020-12-27 (Actual)

PRIMARY OUTCOMES:
Safety- Number of incidents of trial duration above 300 hours | 12 months
  The duration of the study procedures will be no more than 12.5 days
Safety measurments of the C-Scan System regarding SUSAR | 12 months
  No Incidents of SUSAR according to CTCAE scale
Evaluation of the performance of the C-scan System in detecting polyps≥10 mm compared to FIT results | 12 months
  rate of Positive and Negative Agreement of C-Scan System compared to FIT in detecting subjects with polypoid lesions ≥10 mm

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Lewkowicz, Dsc., Study Director — Check-Cap
Locations (4):
- Israel (4):
  - Bnai Zion Medical Center, Haifa, North
  - Rambam Medical Center, Haifa, North
  - Haemek Medical Center, Afula
  - Tel Aviv Sorasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No